CLINICAL TRIAL: NCT04928859
Title: Study on Efficacy and Safety of Human Albumin in Burn Shock Recovery
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-489
Record Dates: First submitted 2021-06-02; First posted 2021-06-16 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2014-06

CONDITIONS: Burns Shock
Keywords: burns; shock; recovery; human albumin; effect
MeSH Terms: conditions — Burns; Shock | interventions — Albumins; Serum Albumin, Human

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- the albumin group: The albumin group, the patients who used albumin for resuscitation during their hospitalization in the burn ward constituted the albumin group.
  Interventions: Drug: Albumin
- the control group: The control group, the patients who did not use albumin during their hospitalization in the burn ward constituted the control group.

INTERVENTIONS:
Drug: Albumin — At least one dose of human albumin was used for the patients during hospitalization in the burn ward consisted the albumin group.
  The patients who have no albumin use during their hospitalization in the burn ward consisted the control group.
  Other Names: human albumin
  Groups: the albumin group

SUMMARY:
To explore the effects and safety of human albumin in burn shock recovery, and then provide a theoretical basis for its rational use.

DETAILED DESCRIPTION:
A retrospective case-control study was conducted. Patients who admitted to the burn ward and needed fluid resuscitation during the period of January 2011 to December 2018 in our unit were identified. Patients were divided into two groups according to the severity of burns, the patients with a 20%<TBSA≤50% constituted the moderate and severe burn group, the patients with a TBSA>50% constituted the severest burn group, and then the patients who used albumin for resuscitation constituted the albumin group, the patients who did not use albumin constituted the control group. The primary outcome was mortality, and the secondary outcomes included hospital stay, ventilator supporting, fluid use, and complications.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* TBSA≥ 20% （TBSA，the total burn area.）
* Admitted to hospital within 24 hours after injury.

Exclusion Criteria:

* STB ≥ 33 μ mol/L
* Cr ≥ 171 μ
* Urine output l< 500 ml / 24 h
* Pregnant and lactating women
* Severe combined injury
* Glucocorticoids users
* Immunosuppressants users
* Patients survived less than 48 hours

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The patients who admitted to the burn ward of the Second Affiliated Hospital, School of Medicine, Zhejiang University and needed fluid resuscitation were identified during the period of January 2011 to December 2018.
Sampling Method: Non-Probability Sample
Enrollment: 364 (Actual)
Dates: Start 2014-06-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
the mortality of the patients | during the patients's hospitalization, an average of 1-2 month.
  The mortality of the patients during their hospitalization.

SECONDARY OUTCOMES:
the length of the patients's hospital stay | during the patients's hospitalization, an average of 1-2 month.
  the Length of the patients's hospital stay,an average of 1-2 month.
the number of patients that using ventilators | during the patients's hospitalization, an average of 1-2 month.
  the number of patients who using ventilators during their hospitalization
Volume of fluid used for resuscitationVolume of fluid used for resuscitation the volume of the patients's resuscitation fluid | during the patients's hospitalization, an average of 1-2 month.
  the volume of the patients's resuscitation fluid using "mL" as the measurement
the number of complications that the patients occurred | during the patients's hospitalization, an average of 1-2 month.
  the number of complications that the patients occurred during their hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Hai-Bin Dai, doctor, Study Director — Second Affiliated Hospital, School of Medicine, Zhejiang University

IPD SHARING:
Plan to Share IPD: No